CLINICAL TRIAL: NCT02231359
Title: Berodual® Respimat® 20/50µg/Dose Solution for Inhalation in Patients With Chronic Obstructive Airways Disease
Brief Title: Berodual® Respimat® Solution for Inhalation in Patients With Chronic Obstructive Airways Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 215.1363
Record Dates: First submitted 2014-09-02; First posted 2014-09-04 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Inhalation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- chronic obstructive airways disease patients
  Interventions: Drug: Berodual® Respimat® solution for inhalation

INTERVENTIONS:
Drug: Berodual® Respimat® solution for inhalation

SUMMARY:
Tolerability, efficacy and handling of Berodual® Respimat® 20/50µg/dose solution for inhalation in patients with chronic obstructive airways disease in daily practice

ELIGIBILITY:
Inclusion Criteria:

* Men and women presenting with the symptoms of chronic obstructive airways disease were given Berodual® Respimat® 20/50µg/dose solution for inhalation only where this was considered necessary in medical terms
* Patients who have not been treated prior to the post-marketing surveillance study as well as patients who have been treated with Berodual® metered dose inhaler (MDI) or other respiratory medications prior to the Post-Marketing Surveillance Study could be included

Exclusion Criteria:

* Patients presenting with the general and specific contraindications listed in the Patient Information Leaflet and the Basic Product Information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diagnosis chronic obstructive airways disease recruited at general practitioners, internal specialists and specialists in pneumology in practice
Sampling Method: Non-Probability Sample
Enrollment: 2006 (Actual)
Dates: Start 2004-01; Primary Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Change in overall severity of clinical picture rated on 3-point scale | up to 12 weeks
Change in breathlessness rated on a 4-point scale | up to 12 weeks
Change in restriction of activity due to breathlessness rated on a 4-point scale | up to 12 weeks
Change in number of awakening due to nocturnal breathlessness rated on 4-point scale | up to 12 weeks
Global assessment of efficacy by the patients rated on 5-point scale | after 4, 8 and 12 weeks
Global assessment of efficacy by the investigator rated on 5-point scale | after 4, 8 and 12 weeks
Number of patients with adverse drug reactions | up to 12 weeks
Assessment of tolerability on a 5-point scale | after 4, 8 and 12 weeks